CLINICAL TRIAL: NCT01560052
Title: Therapeutic Evaluation of Steroids in IgA Nephropathy Global Study Low Dose Study
Brief Title: Therapeutic Evaluation of Steroids in IgA Nephropathy Global Study (TESTING Low Dose Study)
Acronym: TESTING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GI-R-01-2011
Record Dates: First submitted 2012-03-15; First posted 2012-03-21 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: IgA Glomerulonephritis
Keywords: end stage kidney disease; IgA nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA; Kidney Failure, Chronic | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral methylprednisolone (Active Comparator): oral methylprednisolone
  Original Cohort:
  Methylprednisolone group; start at 0.8mg/kg/day with a maximal 48mg/kg/day x 2months, taper by 8mg/day every month with optimal blood pressure control and full dose of ACE inhibitors or ARBs as recommended by guidelines.
  Low Dose Cohort:
  Methylprednisolone group; start at 0.4mg /kg/day with a maximal dose of 32mg/day and a minimum dose of 24mg/day, reducing over 6-9months.
  All participants will also receive standard guideline based care, without steroid therapy. Prophylactic trimethoprim/sulfamethoxazole (a single strength tablet daily or half a double strength tablet daily) will be used during the first 3 months in the low-dose cohort, after randomisation, for the prevention of severe PJP infection, unless there is a documented sulfa allergy.
  Interventions: Drug: methylprednisolone
- placebo (Placebo Comparator): Original Cohort:
  Matching placebo; Optimal blood pressure control and full dose of ACE inhibitors or ARBs as recommended by guidelines; Low Dose Cohort; Matching placebo: Optimal blood pressure control and full dose of ACE inhibitors or ARBs as recommended by guidelines.
  All participants will also receive standard guideline based care, without steroid therapy. Prophylactic trimethoprim/sulfamethoxazole (a single strength tablet daily or half a double strength tablet daily) will be used during the first 3 months in the low-dose cohort, after randomisation, for the prevention of severe PJP infection, unless there is a documented sulfa allergy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: methylprednisolone — Original Cohort:
  Oral methylprednisolone or placebo 0.8mg/kg/day with a maximum of 48mg/day x 2months, taper by 8mg/day every month, patients will also receive optimal blood pressure control and full dose of ACE inhibitors or ARBs as recommended by guidelines
  Low Dose Cohort:
  Oral methylprednisolone or placebo 0.4mg/kg/day with a maximum 32mg/day and minimum of 24mg/day then reducing over 6-9months. All the patients will also receive optimal blood pressure control and full dose of ACE inhibitors or ARBs as recommended by guidelines throughout the trial.
  Prophylactic trimethoprim/sulfamethoxazole (a single strength tablet daily or half a double strength tablet daily) will be used during the first 3 months after randomisation in the low dose cohort, for the prevention of severe PJP infection, unless there is a documented sulfa allergy.
  Other Names: Medrol
  Arms: oral methylprednisolone
Drug: Placebo — Intervention: Drug: Placebo
  Original Cohort:
  Matching placebo tablets, all the patients will receive optimal blood pressure control and full dose of ACE inhibitors or ARBs as recommended by guidelines throughout the trial.
  Low Dose cohort:
  Matching placebo will be given reducing over 6-9months. All the patients will also receive optimal blood pressure control and full dose of ACE inhibitors or ARBs as recommended by guidelines throughout the trial.
  Prophylactic trimethoprim/sulfamethoxazole (a single strength tablet daily or half a double strength tablet daily) will be used during the first 3 months after randomisation in the low dose cohort, for the prevention of severe PJP infection, unless there is a documented sulfa allergy
  Arms: placebo

SUMMARY:
This study will evaluate the long-term efficacy and safety of low dose oral methylprednisolone compared to matching placebo, on a background of routine RAS inhibitor therapy, in preventing kidney events in patients with IgA nephropathy and features suggesting a high risk of progression.

DETAILED DESCRIPTION:
IgA glomerulonephritis is the most common primary glomerulonephritis, and immunosuppression with steroids has been suggested to be a potential protective therapy, although the benefits and risks have not been clearly established.

The TESTING study was established to compare the effects of oral methylprednisolone 0.8 mg/kg/day weaning over 6-8 months, to matching placebo on the risk of kidney failure events, using a double-blind, randomised, controlled design.

After the randomisation of 262 participants to the TESTING an imbalance in serious adverse events was noted between the methylprednisolone and placebo arms of the trial by the Data Monitoring Committee, mostly due to infection. As the data also suggested likely benefit on kidney outcomes, a further 240 participants will be randomised to methylprednisolone 0.4 mg/kg/day compared to matching placebo (The TESTING low-dose group). Oral sulfamethoxazole/trimethoprim will also be provided to reduce the risk of infection All participants will undergo long term follow-up until at least 160 primary outcome events are observed (expected to be an average of at least 4 years), and the effects of steroids on the risk of the composite kidney outcome will be assessed on the study population as a whole, stratified for treatment regimen so long as there is no evidence of significant heterogeneity in the efficacy at reducing the primary outcome.

Each of the original and the low-dose cohorts in TESTING will also have separate power to detect reductions in proteinuria and effects on average eGFR, along with effects on important safety outcomes with the steroid regimens used.

ELIGIBILITY:
Inclusion Criteria:

1. IgA nephropathy proven on renal biopsy.
2. Proteinuria: >=1.0g/day while receiving maximum tolerated dose of RAS blockade following the recommended treatment guidelines of each country where the trial is conducted.
3. eGFR: 30 to 120ml/min per 1.73m²(inclusive) while receiving maximum tolerated RAS blockade

Exclusion Criteria:

1. Indication for immunosuppressive therapy with corticosteroids, such as:

   * Minimal change renal disease with IgA deposits Crescents present in >50% of glomeruli on a renal biopsy within the last 12 months.
2. Contraindication to immunosuppressive therapy with corticosteroids, including:

   * Active infection, including HBV infection or clinical evidence of latent or active tuberculosis (nodules, cavities, tuberculoma, etc)
   * Malignancy within the last 5 years, excluding treated non-melanoma skin cancers (ie. squamous or basal cell carcinoma)
   * Current or planned pregnancy or breastfeeding women of childbearing age who are not able or willing to use adequate contraception.
3. Systemic immunosuppressive therapy in the previous year.
4. Malignant /uncontrolled hypertension (>160mm systolic or 110mmHg diastolic)
5. Current unstable kidney function for other reasons, e.g. macrohaematuria induced acute kidney injury
6. Age <18 years old
7. Secondary IgA nephropathy: e.g. due to lupus, liver cirrhosis, Henoch- Schonlein purpura
8. Patients who are unlikely to comply with the study protocol in the view of the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2012-05-05 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
Progressive kidney failure | 1-6 years
  Progressive kidney failure, which is a composite of a 40% decrease in eGFR, the development of end stage kidney disease defined as a need for maintenance dialysis or kidney transplantation, and death due to kidney disease.
primary outcome for low dose cohort | 1 year
  Change in proteinuria from baseline at 6 and 12 months Mean change in eGFR at 6 and 12 months

SECONDARY OUTCOMES:
The composite of ESKD, 30% decrease in eGFR and all cause death | 1-6 years
The composite of ESKD 40% decrease in eGFR and all cause death | 1-6 years
The composite of ESKD 50% decrease in eGFR and all cause death | 1-6 years
Annual eGFR decline rate | 1-6 years
Each ESKD , death due to kidney disease and all cause death | 1-6 years
Time averaged proteinuria post-randomisation | 1-6 years

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, Principal Investigator — Peking University; Vlado Perkovic, Principal Investigator — The George Institute
Locations (66):
- Australia (5):
  - Concord Repatriation and General Hospital, Concord, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Melbourne, Victoria
- Canada (8):
  - University of Calgary/Alberta Health Services, Calgary, Alberta
  - University of Alberta Hospitals, Edmonton, Alberta
  - St Pauls Hospital, Vancouver, British Columbia
  - St. Joseph's Healthcare, Hamiliton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto General Hospital,, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
- China (40):
  - Chinese PLA General Hospital (301 Hospital), Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - ongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital, Wuhan University, Wuhan, Hubei
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technology,, Baotou, Inner Mongolia
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia
  - General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Jilin Province FAW General Hospital [Jilin University Fourth Hospital], Changchun, Jilin
  - he First Affiliated Hospital of Dalian Medical University, Dalian, Dalian, Liaoning
  - Shengjing Hospital Of China Medical University, Shengyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The First Affiliated Hospital of Shangdong First Medical University,Shangdong Provincial Qianfoshin, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Jinan Military General Hospital, Jinan, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - he Second Hospital of Shanxi Medical University, Taiyuan, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Academy of Medical Science, Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital, Zhejiang University of Medicine, Hangzhou, Zhejiang
  - Hangzhou Hospital of Traditional Chinese Medicine,, Hangzhou, Zhejiang
  - Ningbo Urology & Nephrology Hospital, Ningbo, Zhejiang
  - Zhejiang Provincial People's Hospital, Sangzhou, Zhejiang
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - XinQiao Hospital, Third Military Medical University, Chongqing
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Ruijin Hospital, Shanghai Jiaotong University, School of Medicine, Shanghai
  - Huashan Hospital, Medical Centre of Fudan University, Shanghai
- Princess Margaret Hospital, Kowloon, Hong Kong
- India (6):
  - Osmania General Hospital, Hyderabad, Andhra Pradesh
  - Nizam's Institute of Medical Science, Hyderabad, Andhra Pradesh
  - Calicut Medical College, Kozhikode, Kerala
  - Post Graduate Institue of Medical Education and Reasearch, Chandigarh, Punjab
  - Madras Medical College, Chen, Tamil Nadu
  - Sanjay Gandhi Post Graduate Institute of Medical Science, Lucknow, Uttar Pradesh
- Malaysia (6):
  - Hospital Sultanah Aminah, Johor Bahru, Johor
  - Hospital Kuala Lumpur, Kuala Lumpur, Kulala Lumpur
  - Hospital Tuanku Jaafar Seremban, Seremban, Negri Seremban
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Umum Sarawak, Kuching, Samarahan
  - University Malaysia Medical Centre, Kuala Lumpur

REFERENCES:
- [Derived] Xu LL, Zhou XJ, Bi W, Zhang P, Shi SF, Liu LJ, Lv JC, Zhang H. Genetic Determinants of Steroid Responsiveness in IgA Nephropathy. J Am Soc Nephrol. 2025 Dec 11. doi: 10.1681/ASN.0000000977. Online ahead of print. No abstract available. PMID 41563292
- [Derived] Lv J, Wong MG, Hladunewich MA, Jha V, Hooi LS, Monaghan H, Zhao M, Barbour S, Jardine MJ, Reich HN, Cattran D, Glassock R, Levin A, Wheeler DC, Woodward M, Billot L, Stepien S, Rogers K, Chan TM, Liu ZH, Johnson DW, Cass A, Feehally J, Floege J, Remuzzi G, Wu Y, Agarwal R, Zhang H, Perkovic V; TESTING Study Group. Effect of Oral Methylprednisolone on Decline in Kidney Function or Kidney Failure in Patients With IgA Nephropathy: The TESTING Randomized Clinical Trial. JAMA. 2022 May 17;327(19):1888-1898. doi: 10.1001/jama.2022.5368. PMID 35579642
- [Derived] Lv J, Zhang H, Wong MG, Jardine MJ, Hladunewich M, Jha V, Monaghan H, Zhao M, Barbour S, Reich H, Cattran D, Glassock R, Levin A, Wheeler D, Woodward M, Billot L, Chan TM, Liu ZH, Johnson DW, Cass A, Feehally J, Floege J, Remuzzi G, Wu Y, Agarwal R, Wang HY, Perkovic V; TESTING Study Group. Effect of Oral Methylprednisolone on Clinical Outcomes in Patients With IgA Nephropathy: The TESTING Randomized Clinical Trial. JAMA. 2017 Aug 1;318(5):432-442. doi: 10.1001/jama.2017.9362. PMID 28763548
- [Derived] Yeo SC, Liew A, Barratt J. Emerging therapies in immunoglobulin A nephropathy. Nephrology (Carlton). 2015 Nov;20(11):788-800. doi: 10.1111/nep.12527. PMID 26032537